CLINICAL TRIAL: NCT06533891
Title: Effects of Omega-3 Fatty Acid Supplementation and Physical Training on Metabolic Health
Acronym: EXC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Supplements expired during COVID shutdown
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ann Skulas-Ray, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1912251764
Record Dates: First submitted 2020-02-03; First posted 2024-08-01 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DPA enriched n-3 (Experimental): 4 g/d DPA enriched n-3 concentrate (~980 mg DPA, 380 mg EPA, 1720 mg DHA)
  Interventions: Dietary Supplement: DPA enriched n-3
- n-3 control (Active Comparator): 4 g/d n-3 control (~980 oleic acid, 380 mg EPA, 1720 mg DHA)
  Interventions: Dietary Supplement: n-3 control
- Placebo (Placebo Comparator): 4 g/d placebo control ("light" olive oil)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DPA enriched n-3 — 4 g/d DPA enriched n-3 concentrate (~980 mg DPA, 380 mg EPA, 1720 mg DHA)
  Arms: DPA enriched n-3
Dietary Supplement: n-3 control — 4 g/d n-3 control (~980 oleic acid, 380 mg EPA, 1720 mg DHA)
  Arms: n-3 control
Dietary Supplement: Placebo — 4 g/d placebo control ("light" olive oil)
  Arms: Placebo

SUMMARY:
The degree of insulin resistance in an individual can be monitored by several means including blood concentrations of insulin, triglycerides, HDL-C, and eventually glucose. In particular, the ratio of triglycerides to HDL-C reflects the severity of insulin resistance's impact on liver-mediated lipoprotein transport and may be a sensitive measure of early insulin resistance when fasting glucose levels are still in the normal range (compensated by higher output of insulin). High triglycerides and low HDL-C indicate poor metabolic health and increased risk of fatty liver and atherosclerotic cardiovascular diseases.

Two diet and lifestyle strategies that have shown therapeutic promise are 1) supplementation with omega-3 fatty acids and 2) aerobic exercise training. Omega-3 fatty acids can prevent the development of insulin resistance but have not been successful in reversing established insulin resistance. Importantly, omega-3 fatty acids are effective for improving the ratio of triglycerides to HDL-C in blood and reducing the amount of fat in the liver. Aerobic exercise has demonstrated greater success for reversing established insulin resistance, but it is not known if and to what degree supplementation with omega-3 fatty acids could potentiate its therapeutic efficacy and vice versa regarding dyslipidemia. Both omega-3 fatty acids and exercise lead to increased blood concentrations of beneficial oxygenated lipid compounds (termed oxylipins) that regulate inflammatory and metabolic processes (including insulin resistance) linked to the development of NAFL.

In preparation for studies of people in poorer metabolic health, the investigators will conduct a pilot and feasibility study of relatively inactive younger adults with low dietary intake of omega-3 fatty acids to assess whether increased aerobic physical activity combined with omega-3 supplementation leads to greater improvements in blood concentrations of triglycerides, HDL-C, and their ratio, as well as concentrations of oxylipins in the blood. The investigators will also assess whether a less studied omega-3 fatty acid, called DPA, may have effects above and beyond those conferred by EPA and DHA (which are concentrated in prescription omega-3 fatty acid products).

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled clinical study. The treatment phase will span a continuous 6-week period. Prior to the treatment phase, participants will be assigned to receive the DPA enriched n-3 supplement, conventional n-3 supplement, or identical placebo. A computer program will be used to randomly assign participants to a treatment group.

Intervention protocol and study treatments:

Study capsules will be provided tri-weekly at the Food, Bioactives, & Health Lab on the University of Arizona campus. Participants may schedule pick-up times that are most suitable for their schedules. A staff member will be available to meet with participants at each tri-weekly pick-up appointment.

The treatments are as follows:

* 4 g/d DPA enriched n-3 concentrate (~980 mg DPA, 380 mg EPA, 1720 mg DHA)
* 4 g/d n-3 control (~980 oleic acid, 380 mg EPA, 1720 mg DHA)
* 4 g/d placebo control ("light" olive oil)

During the 6-week treatment phase, participants will consume 4 g/day of the DPA-enriched concentrate, n-3 matched control, or placebo control. Participants will be required to avoid consuming any other food or supplements that contain n-3 FA during treatment phases. They will also be asked to engage in exercise ad libitum while wearing a heart rate monitor for the 6-week period.

The supplementation period will be at least 6 weeks in length. However, it can be extended by 3 weeks (up to 9 weeks total) to accommodate scheduling challenges due to illness, travel, etc. For example, should a participant be unable to come in on two separate mornings for testing after 6 weeks of supplementation, they may continue the supplement and schedule testing for the following week.

Screening:

Potential participants will be interviewed by telephone to determine their initial eligibility. If they remain eligible after the telephone screening, they will be further screened at the Food, Bioactives, & Health Lab. This screening visit will consist of: filling out forms (informed consent, medical history, personal information); measuring height and weight so body mass index (BMI) can be calculated; and measuring blood pressure (BP). If it is determined that they are still eligible following these measurements, a blood sample will be taken and a complete blood cell count, health panel including liver and kidney function, and a blood fat panel will be performed (approximately 15 mL of blood or ~1 tablespoon will be taken). If the initial blood draw is unsuccessful, it may need to be repeated, with permission of the participant. Females of child-bearing age will be given a urine pregnancy test. Study investigators will review all of the screening data. Participants meeting eligibility criteria will be scheduled for baseline data collection and supplementation will begin thereafter.

• Urine Pregnancy Testing: Female participants of childbearing age will be asked to provide a urine sample for pregnancy testing at baseline. If a participant is pregnant, she will not be able to participate in the study.

Baseline and endpoint visits (3 total):

Participants will undergo additional clinical and anthropometric assessments for one day at baseline (screening values will be used as the second measure) and two days for endpoint visits (at the end of the 6-week treatment phase). The baseline visit will be scheduled within 2 weeks of the participant's screening visit. Participants will be required to fast overnight (12 hours with no food or drink except water) and abstain from alcohol for 48 hours prior to each testing day. To ensure participant eligibility, a brief assessment will be administered. If a participant does not meet the requirements, their visit will be rescheduled. Testing will be conducted at the Food, Bioactives, & Health Lab and the procedures are described in more detail below.

• Blood Sampling: Prior to having their blood taken, participants will be asked not to consume any food or drink except water for 12 hours and to avoid alcohol for 48 hours. Participants also should not engage in vigorous physical activity for 12 hours prior to having their blood taken. Two blood samples will be taken at baseline and at the end of the treatment phase (for a total of 3 times after eligibility screening). On two separate days, a blood sample will be taken from the participant's arm after a 12-hour fast (no food or drink except water). If the initial blood draw is unsuccessful it may need to be repeated, with the participant's permission. Approximately 60 mL (4 tablespoons) of blood will be collected at baseline and at the end of each treatment phase, over two days separated by at least 24 hours. This will be collected as ~52 mL on one day and ~7.5 mL on the other day. Throughout the entire study, blood will be taken 4 times for a total amount of ~130 mL (~8.5 tablespoons), including the blood taken for screening tests prior to the start of the study (~15 mL or 1 tablespoon).

* At the end of the testing period, blood will be tested for the following: glucose, insulin, triglycerides, HDL-C, non-HDL-C, and concentrations of inflammatory markers. Red blood cell fatty acid concentrations will also be measured to assess compliance.
* On an additional day at the end of each testing period, participants will provide a blood sample (~7.5 mL) to repeat lipid measurements, which can vary day-to-day.

Blood samples will be stored and analyzed after all participants have completed the study. Study results will be available after study completion (which may take 2 years or longer).

* Rockport Walking Test: VO2 max will be calculated using the Rockport Walking Test. The test will be conducted using the indoor track at the Rec Center. Participants will be allowed to warm-up and stretch prior to starting the test, and will then walk 1 mile as quickly as they are able. Finishing times will be noted, and heart rate will be measured for 15 seconds immediately after.
* Body Composition Assessment: Body composition will be determined using a 4-point bioelectrical impedance analysis device. Weight and waist circumference will also be measured.

Ad Libitum Physical Training: Participants will be asked to engage in physical training ad libitum during the 6-week study period. Participants will be granted access to the Rec Center and all Rec Center group fitness classes. During the first week of training, participants will work with a qualified study intern to establish a physical activity baseline and initial exercise plan. Participants will meet with their study intern intermittently after the first week to aid in adherence to safe practices and study procedures.

Midpoint Visits: Supplements will be provided every 3 weeks at the Food, Bioactives, and Health Lab on the University of Arizona campus. Participants may schedule pick up times that work best with their schedule. A study staff member will be available at each pick up visit to meet with participants to answer questions or discuss side effects.

ELIGIBILITY:
Inclusion Criteria:

* Light to moderate activity level
* BMI of 18-29 kg/m2
* Consistent dosage for any medication/supplements taken for inflammatory conditions
* Ability to abstain from alcohol for 48 hours prior to lab testing
* Low fish consumption (<2 serving/week), no use of omega-3 or fish oil supplements

Exclusion Criteria:

* Pregnant or lactating
* Use of medications for blood thinning, elevated lipids, blood pressure, or glucose
* Allergy to fish
* Any condition for which exercise is contraindicated
* Intolerance to physical training

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Triglyceride/HDL-C ratio | 6 weeks
  Triglyceride/HDL-C ratio

OTHER OUTCOMES:
Oxylipins | 6 weeks
  Concentrations of specific omega-3 derived pro-resolving lipid mediators
Glucose | 6 weeks
  Glucose
C-reactive protein (CRP) | 6 weeks
  C-reactive protein (CRP)
Insulin | 6 weeks
  Insulin
VO2 max | 6 weeks
  VO2 max
Weight | 6 weeks
  Weight
Waist circumference | 6 weeks
  Waist circumference
Body fat percentage | 6 weeks
  Body fat percentage

IPD SHARING:
Plan to Share IPD: No